CLINICAL TRIAL: NCT00854412
Title: The Effect of Weight Loss on Serum Mannose-Binding Lectin (MBL) Levels
Brief Title: The Effect of Weight Loss on Serum Mannose-Binding Lectin(MBL) Levels
Acronym: WLMBL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Pernille Høyem MD, PhD-student, Medical Department M, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MBL1
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Obesity; Weight Loss
Keywords: Obesity; Weight loss; Very low-calorie diet; Mannose-binding lectin; Insulin resistance
MeSH Terms: conditions — Obesity; Weight Loss; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Weight loss — Very low-calorie diet (VLCD) of 800 kcal/day for 8 weeks

SUMMARY:
High levels of mannose-binding lectin (MBL), an activator of a part of the immune system called the complement system, have been associated with increased mortality and risk of early signs of kidney damage in patients with type 2 diabetes. The effect of weight loss and changes in insulin resistance on MBL levels have been poorly elucidated.

This study includes 36 nondiabetic obese subjects, who will receive a very low- calorie diet (VLCD) of 800 kcal/day for 8 weeks.

Fasting blood samples will be obtained at baseline and after 8 weeks of VLCD and concentrations of MBL, glucose and insulin will be measured. Insulin resistance is assessed using the HOMA-IR method.

ELIGIBILITY:
Inclusion Criteria:

* Obese

Exclusion Criteria:

* Diabetes
* Other severe disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 1995-03; Primary Completion 1995-06 (Actual); Study Completion 1995-06 (Actual)